CLINICAL TRIAL: NCT06119893
Title: Effect of Submucosal Dexamethasone on Postoperative Pain, Swelling and Trismus After Periodontal Surgery: Randomized Clinical Study
Brief Title: The Use of Submucosal Dexamethasone After Periodontal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Dicle Altındal, DDS, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13.07.2021/08
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Pocket; Pain; Swelling/ Edema; Patient Satisfaction; Periodontitis
Keywords: pain; dexamethasone; surgical flaps
MeSH Terms: conditions — Periodontal Pocket; Pain; Edema; Patient Satisfaction; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patient received an indication periodontal flap surgery. In this randomized controlled split mouth study, the patient underwents periodontal flap surgery in their mandibular. Following local anesthesia (2% lidocaine and 1:100,000 epinephrine), sulcular incisions were made. Vertical incision was not used in any operation. The mucoperiosteal flap was elevated until the buccal and lingual bone defects were adequately exposed. Defects were thoroughly debrided firstly by using periodontal curettes, and then cleaned by piezoelectric ultrasonic scaler to ensure all granulation tissues were thoroughly removed. Buccal and lingual flaps were closed primarily. In the control group, 2 mL 0.9% isotonic sodium chloride (saline) with 27-gauge single-type disposable syringes was applied to the buccal surface of flap after the operation
  Interventions: Drug: submucosal 2 mL 0.9% isotonic sodium chloride application
- Test Group (Active Comparator): Patient received an indication periodontal flap surgery. In this randomized controlled split mouth study, the patient underwents periodontal flap surgery in their mandibular. Following local anesthesia (2% lidocaine and 1:100,000 epinephrine), sulcular incisions were made. Vertical incision was not used in any operation. The mucoperiosteal flap was elevated until the buccal and lingual bone defects were adequately exposed. Defects were thoroughly debrided firstly by using periodontal curettes, and then cleaned by piezoelectric ultrasonic scaler to ensure all granulation tissues were thoroughly removed. Buccal and lingual flaps were closed primarily. In the test group, 8 mg (2 mL) submucosal dexamethasone with 27-gauge single-type disposable syringes was applied to the buccal surface of flap after the operation
  Interventions: Drug: submucosal 8 mg (2 mL) dexamethasone application

INTERVENTIONS:
Drug: submucosal 8 mg (2 mL) dexamethasone application — The mucoperiosteal flap was applied. After operation, submucosal dexamethasone 8 mg (2 mL) was applied to the operation area as a test group.
  Other Names: Periodontal flap surgery
  Arms: Test Group
Drug: submucosal 2 mL 0.9% isotonic sodium chloride application — The mucoperiosteal flap was applied. After operation, 2 mL 0.9% isotonic sodium chloride was applied to the operation area as a control group
  Other Names: Periodontal flap surgery
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of submucosal 8 mg (2 mL) dexamethasone on postoperative pain, swelling, chewing efficiency, trismus, healing, and discomfort after periodontal flap surgery

DETAILED DESCRIPTION:
Periodontitis is an oral inflamatuar disease caused by specific microorganisms, is characterized by attachment loss, alveolar bone resorption, pathological pocket formation. This disease causes deep periodontal pockets associated with deep intrabony defects as well as various clinical problems. For management overcome these problems, various approaches have been proposed in the treatment of periodontitis, including initial periodontal treatment such as scaling and root planing, followed by flap surgery, resective bone surgery and periodontal regeneration when applicable. However, periodontal flap surgery applied in these approaches causes undesirable side effects such as pain and swelling. To overcome these disorders, studies continue to investigate by using various medication regimens include pre, intra or post operative drugs.

Dexamethasone is a synthetic steroidal anti-inflammatory drug used to control pain, swelling, and inflammation occurring in third molar surgeries, periodontal therapy and periodontal surgeries, implant surgery, and endodontic treatment. In the literature, dexamethasone application is frequently used in oral surgery before or after third molar tooth extraction. There is limited research on dexamethasone applications in periodontal flap surgery. lt has been evaluated the effectiveness of oral use of etoricoxib and dexamethasone in preventing pain after open flap debridement surgery. Some authors used 4 mg dexamethasone tablets before mucoperiosteal flap surgery and reported that the pain level in the dexamethasone group was lower than placebo at the 3rd hour. It has been reported positive results where preferred its use intravenously in the postoperative management of periodontal surgery. However, to the investigators knowledge, there is no study in the literature in which dexamethasone is applied submucosally after periodontal flap surgery. Accordingly, the hypothesis of this study was that submucosal application of dexamethasone in periodontal flap surgery would have a positive effect on pain and patient comfort. In light of all these scientific data, this study aimed to evaluate the effect of submucosal dexamethasone application periodontal flap surgery on postoperative pain, swelling, chewing efficiency, trismus, healing and discomfort.

ELIGIBILITY:
Inclusion Criteria:

1. pocket depth ≥5mm;
2. systemically healthy;
3. without drug allergy;
4. without any blood disease;
5. not using medication (anti-platelet, anticoagulant, immunosuppressant medication);
6. received no any periodontal surgery in the last 6 months;

Exclusion Criteria:

1. poor oral hygiene;
2. smoking;
3. any systemic disease that would affect the surgical operation;
4. problem with the kidneys or adrenal glands;
5. connective tissue disease or immunodeficiency;
6. breastfeeding period or pregnancy.
7. high dental anxiety

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
VAS | Every hour for the first 8 hours on the first day of the operation, and three times a day on the 2nd, 3rd, 4th and 7th days
  Visual analogue scale (VAS) was assessed to monitor the degree of pain.VAS is a scale that rates pain severity from 0 to 10. (0 = no pain to 10 = severe pain),
NRS-101 | Every hour for the first 8 hours on the first day of the operation, and three times a day on the 2nd, 3rd, 4th and 7th days
  101-point numeric rate scale (NRS-101) was assessed to monitor the degree of pain. NRS-101 is a 101-point numerical ratio scale that rates pain severity from 0 to 100. (0 = no pain to 100 = severe pain),
Swelling | Patients were evaluated for swelling on the preoperative, the1st, 2nd, and 7th days after the operation
  Linear measurements were taken for swelling with a millimeter tape measure. Measurements were made between the angle of the mandible and the mentus, labial commissure, nasal ala, outer corner of the eye and tragus. The average of these five measurements was noted.

SECONDARY OUTCOMES:
Trismus | It was evaluated for trismus on the preoperative, the 1st, 2nd, and 7th days after the operation
  For trismus evaluation, mouth opening was measured using a millimetric ruler by measuring the distance between the mesial-incisal corners of the upper right and lower right central incisors at the maximum jaw opening while the patient was sitting upright.
Chewing efficiency | It was evaluated for chewing efficiency on the 1st, 2nd, and 7th days after the operation
  Chewing efficiency was scored by the patients as 1) very poor, 2) poor, 3) good, 4) very good and 5) excellent.
Healing of operation area | It was evaluated for healing of operation area on the 1st, 2nd, and 7th days after the operation
  Healing at the operative site in terms of infection was scored by clinician as follows: 1) very poor, 2) poor, 3) good, 4) very good, and 5) excellent healing
Discomfort | It was evaluated for discomfort on the 1st, 2nd, and 7th days after the operation
  In the evaluation of discomfort, the four-point verbal rating scale (VRS-4) and a questionnaire questioning patient comfort were used. The questionnaire was scored with this four-point scoring system (Pain in this scoring: 1) none, 2) mild, 3) moderate, 4) severe).
Analgesics consumed | The number of analgesics used each day during the first 7 days was noted by the patient in the pain diary
  The number of analgesics used was noted by the patient in the pain diary.
General satisfaction | 14th day after operation
  On the day of removing suture, the patients' general satisfaction levels were measured with a 5-point scale ( 1) poor, 2) reasonable, 3) good, 4) very good and 5) excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Dicle Altindal, DDS, Principal Investigator — Yuzuncu Yil University; Anas ALSAFADI, PhD, Study Chair — Special dental clinic; Basem ALSHUJAA, PhD, Study Chair — Special dental clinic; Ahmet Cemil Talmac, PhD, Study Chair — Yuzuncu Yil University; Bilal Ege, PhD, Study Chair — Adiyaman University; Metin Calisir, PhD, Study Chair — Adiyaman University; Nazli Zeynep Alpaslan, PhD, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vieth MP, Deas DE, Archontia Palaiologou A, Diogenes A, Mader MJ, Mealey BL. Effect of intravenous dexamethasone on postoperative pain and swelling following periodontal flap surgery: A randomized controlled trial of patient-centered outcomes. J Periodontol. 2022 Feb;93(2):237-245. doi: 10.1002/JPER.21-0153. Epub 2021 Jun 3. PMID 34021915
- [Background] Steffens JP, Santos FA, Pilatti GL. Postoperative periodontal pain prevention using two dexamethasone medication protocols: a double-blind, parallel-group, placebo-controlled randomized clinical trial. Am J Dent. 2011 Dec;24(6):354-6. PMID 22263332
- [Background] Aksoy F, Ege B. The effect of pretreatment submucosal injections of tramadol and dexamethasone on post-endodontic pain in mandibular molar teeth with symptomatic irreversible pulpitis: a randomized controlled clinical trial. Int Endod J. 2020 Feb;53(2):176-185. doi: 10.1111/iej.13246. Epub 2019 Nov 28. PMID 31702056
- [Derived] Altindal D, Alsafadi A, Alshujaa B, Talmac AC, Ege B, Calisir M, Alpaslan NZ. Effect of submucosal dexamethasone on postoperative pain, swelling and trismus after periodontal surgery: a randomized clinical study. Clin Oral Investig. 2024 Dec 4;28(12):681. doi: 10.1007/s00784-024-06076-5. PMID 39627624